CLINICAL TRIAL: NCT05842902
Title: Pilot Trial Testing Mobile Health Psychosocial Intervention for Adolescents and Young Adults With Cancer
Brief Title: Resilience Mobile App for Teens and Young Adults With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Nancy, Assistant Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004006
Record Dates: First submitted 2023-04-21; First posted 2023-05-06 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: Mobile health; Quality of life; Adolescent; Young Adult; Psychosocial factors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized waitlist design: AYAs will be randomized 1:1 to psychosocial Usual Care (UC) or UC plus mPRISM. mPRISM will be provided to UC arm at 3-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mPRISM (Experimental): The Experimental (mPRISM) arm will receive mPRISM upon completion of their baseline study surveys.
  Interventions: Behavioral: mPRISM
- Waitlist control (Other): Usual Care (UC) available to both study arms consists of standard non-directed supportive care provided for all patients including an assigned social worker throughout cancer treatment. In a waitlist design, the UC arm will receive mPRISM upon completion of 3-month follow-up surveys.
  Interventions: Behavioral: mPRISM

INTERVENTIONS:
Behavioral: mPRISM — PRISM is a brief, 1:1, skills-based resilience intervention delivered in-person by trained layperson coaches. PRISM's development was based on iterative research within the AYA oncology population, stress and coping theory, resilience theory, and successful cognitive-behavioral and mindfulness interventions. mPRISM is a digital version of the PRISM program with no in-person delivery. mPRISM includes coping skills modules: managing stress, goal-setting, cognitive reframing, and meaning-making.

SUMMARY:
The goal of this pilot trial is to examine whether a mobile app version of the Promoting Resilience in Stress Management (PRISM) intervention is acceptable, easy to use, and helps improve quality of life and mental health symptoms.

DETAILED DESCRIPTION:
Adolescents and Young Adults (AYAs) with cancer are at risk of distress, anxiety, depression, and poor quality of life. The use of mobile applications for psychosocial symptom self-management is appealing to this demographic population but this has not yet been developed and tested.

PRISM is a novel, brief, evidence-based 1:1 intervention that teaches stress management, goal-setting, meaning making, cognitive-behavioral, and mindfulness strategies. Here, we propose to test a mobile health (mHealth) version of PRISM, mPRISM. In a pilot randomized controlled trial, we will evaluate the feasibility, acceptability, and exploratory efficacy of mPRISM using a waitlist control design.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-25 years
* Diagnosis of new malignancy within 12 months of enrollment treated with chemotherapy and/or radiation therapy at Seattle Children's Hospital (SCH)
* Patient able to speak/read/write English or Spanish language
* Cognitively able to participate in mHealth psychosocial intervention and interactive interviews

Exclusion Criteria:

* Patient refusal to participate (any age), or parental refusal to participate for patients less than 18 years of age
* Patients with diagnosis of malignancy >12 months
* Patients with relapsed, recurrent, or refractory disease
* Patient without chemotherapy and/or radiation therapy as part of cancer treatment (e.g., surgical resection only patients are not-eligible)
* Cognitively or physically unable to participate in mHealth psychosocial intervention and surveys

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability of intervention | immediately post-intervention
  The Acceptability of Intervention Measure (AIM) is a well-validated 4-item scale that measures the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. Scale ranges from 4 to 20; higher scores are better.
Appropriateness of intervention | immediately post-intervention
  The Intervention Appropriateness Measure (IAM) is a well-validated 4-item scale that measures the perceived fit, relevance, or compatibility of the innovation or evidence-based practice for a given practice setting, provider, or consumer, and/or perceived fit of the innovation to address a particular issue or problem. Scale ranges from 4 to 20; higher scores are better.
Feasibility of intervention | immediately post-intervention
  The Feasibility of Intervention Measure (FIM) is a well-validated 4-item scale that measures the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Scale ranges from 4 to 20; higher scores are better.

SECONDARY OUTCOMES:
Usability of intervention | immediately post-intervention
  The System Usability Scale (SUS) is a well-validated and widely used 10-item scale to evaluate the perceived usability of digital interventions. Items are rated on a 5-point Likert scale for a total score ranging from 0-100, and scores ≥70 considered adequate usability.
Change in health-related quality of life | immediately post-intervention, 3 months post-intervention
  The PedsQL 4.0 Generic and 3.0 Cancer Module include 50 items evaluating health-related quality of life (HRQOL) of AYAs with cancer. Queries assess physical, emotional, social, and school well-being, plus cancer-related pain and hurt, nausea, procedural anxiety, treatment anxiety, worry, cognitive problems, perceived physical appearance, and communication. Scores are linearly transformed to a 0-100 scale, with higher scores indicating better HRQOL.
Change in resilience | immediately post-intervention, 3 months post-intervention
  The CD-RISC is a well-validated and widely used 10-item instrument to measure inherent resiliency. Questions revolve around personal problem-solving and approaches to adversity. Scores range from 0-40, with higher scores indicating higher resilience.
Change in distress | immediately post-intervention, 3 months post-intervention
  This 6-item scale measures "level of psychological distress experienced in the past month." The instrument strongly discriminates between community cases and non-cases of Diagnostic and Statistical Manual of Mental Disorder (DSM)-V psychiatric disorders such as serious emotional distress or serious mental illness. Scores range from 0-24, with higher scores indicating higher distress.
Change in anxiety and depression | immediately post-intervention, 3 months post-intervention
  7 items assess symptoms of anxiety and depression, respectively, in patients with serious illness. It has been validated in AYAs with chronic illness and cancer survivors, with excellent reliability (α=0.83-0.82). Items are scored 0-3 (subscale range 0-21), with scores ≥8 categorized as borderline abnormal, and ≥11 categorized as abnormal.

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lau N, Palermo TM, Zhou C, Badillo I, Hong S, Aalfs H, Yi-Frazier JP, McCauley E, Chow EJ, Weiner BJ, Ben-Zeev D, Rosenberg AR. Mobile App Promoting Resilience in Stress Management for Adolescents and Young Adults With Cancer: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2024 Jul 30;13:e57950. doi: 10.2196/57950. PMID 39079108